CLINICAL TRIAL: NCT03700944
Title: The Effects of Yoga Training on Rhinitis Symptoms and Cytokines in Allergic Rhinitis Patients
Brief Title: Yoga Training in Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Lecturer, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC 1
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Yoga; Cytokines; Rhinitis symptoms
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Twenty-seven allergic rhinitis patients, aged 18-45 year old, were randomized into 2 groups: control group (CON; n=14) and yoga group (YOG; n=13). The control group had normal life and the yoga group was required to complete protocol with yoga training for a period of 8 weeks, 60 minutes, 3 times a week. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-test and post-test.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YOG (Experimental): The yoga group (YOG) was required to complete protocol with yoga training for a period of 8 weeks, 60 minutes, 3 times a week
  Interventions: Other: Yoga training
- CON (No Intervention): The control group (CON) had normal life.

INTERVENTIONS:
Other: Yoga training — Complete protocol with yoga training for a period of 8 weeks, 60 minutes, 3 times a week.
  Arms: YOG

SUMMARY:
The purpose of this study was to investigate effects of yoga training on rhinitis symptoms and cytokines in allergic rhinitis patients. Twenty-seven allergic rhinitis patients, aged 18-45 year old, were randomized into 2 groups: control group (CON; n=14) and yoga group (YOG; n=13). The control group had normal life and the yoga group was required to complete protocol with yoga training for a period of 8 weeks, 60 minutes, 3 times a week. Physiological variables, lung function variables, allergic rhinitis symptoms variables, and cytokines level in nasal secretion variables were analyzed during pre-test and post-test. The dependent variables between pre-test and post-test were analyzed by a paired t-test. The dependent variables between groups were analyzed by independent t-test. One way repeated measures ANOVA was used to compare the variables among pre-test, after 4 weeks, and after 8 weeks. Differences were considered to be significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of allergic rhinitis diseases
* Clinical symptoms of persistent rhinitis (nasal congestion, sneeze, nasal itching, and running nose) for more than 4 days per week.
* Positive skin prick test (wheal diameter>3 mm.) to house dust mite (D. pteronyssinus) and using normal saline as the negative control.
* Stopped taking all medicine before the study such as antihistamine for at least 3 days, oral steroid and nasal steroid for at least 2 weeks and luekotriene receptor antagonist for at least a week prior to the study, but the patients could take pseudo ephedrine.
* Subjects were not to have participated in a regular exercise program for at least 6 months prior to the start of the study, and to avoid taking any form of dietary supplement during the course of the study.

Exclusion Criteria:

* Asthma
* Chronic rhino-sinusitis
* Hypertension
* Cardiovascular diseases
* A smoking habit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores | 10 minutes
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before and after yoga training protocol. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)

SECONDARY OUTCOMES:
Cytokine in nasal secretion | 10 Minutes
  Nasal secretions collection was performed bilaterally with filter paper strips (7x30 mm Whatman No.42, Whatman, Clifton, NJ). Three filter paper strips were sequentially placed on each anterior portion of the inferior turbinate for 10 min. This filter paper strips were collected into appropriate tubes and centrifuged at 3,000 rpm for 5 min at 4 °C and immediately frozen at -70 °C until later analysis.The levels of cytokines were determined by using Sandwich ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Result] Caggiano S, Cutrera R, Di Marco A, Turchetta A. Exercise-Induced Bronchospasm and Allergy. Front Pediatr. 2017 Jun 8;5:131. doi: 10.3389/fped.2017.00131. eCollection 2017. PMID 28642859
- [Result] Cheema BS, Houridis A, Busch L, Raschke-Cheema V, Melville GW, Marshall PW, Chang D, Machliss B, Lonsdale C, Bowman J, Colagiuri B. Effect of an office worksite-based yoga program on heart rate variability: outcomes of a randomized controlled trial. BMC Complement Altern Med. 2013 Apr 10;13:82. doi: 10.1186/1472-6882-13-82. PMID 23574691
- [Result] Tongtako W, Klaewsongkram J, Jaronsukwimal N, Buranapraditkun S, Mickleborough TD, Suksom D. The effect of acute exhaustive and moderate intensity exercises on nasal cytokine secretion and clinical symptoms in allergic rhinitis patients. Asian Pac J Allergy Immunol. 2012 Sep;30(3):185-92. PMID 23156847
- [Result] Teixeira RUF, Zappelini CEM, Alves FS, da Costa EA. Peak nasal inspiratory flow evaluation as an objective method of measuring nasal airflow. Braz J Otorhinolaryngol. 2011 Jul-Aug;77(4):473-480. doi: 10.1590/S1808-86942011000400011. PMID 21860974
- [Result] Yadav RK, Magan D, Mehta N, Sharma R, Mahapatra SC. Efficacy of a short-term yoga-based lifestyle intervention in reducing stress and inflammation: preliminary results. J Altern Complement Med. 2012 Jul;18(7):662-7. doi: 10.1089/acm.2011.0265. PMID 22830969
- [Result] Zhao N, Liu HJ, Sun YY, Li YZ. Role of interleukin-6 polymorphisms in the development of allergic rhinitis. Genet Mol Res. 2016 Jan 8;15(1). doi: 10.4238/gmr.15016987. PMID 26909898
- [Result] Vijayaraghava A, Doreswamy V, Narasipur OS, Kunnavil R, Srinivasamurthy N. Effect of Yoga Practice on Levels of Inflammatory Markers After Moderate and Strenuous Exercise. J Clin Diagn Res. 2015 Jun;9(6):CC08-12. doi: 10.7860/JCDR/2015/12851.6021. Epub 2015 Jun 1. PMID 26266115
- [Result] Rajbhoj PH, Shete SU, Verma A, Bhogal RS. Effect of yoga module on pro-inflammatory and anti-inflammatory cytokines in industrial workers of lonavla: a randomized controlled trial. J Clin Diagn Res. 2015 Feb;9(2):CC01-5. doi: 10.7860/JCDR/2015/11426.5551. Epub 2015 Feb 1. PMID 25859450
- [Result] Netam R, Yadav RK, Khadgawat R, Sarvottam K, Yadav R. Interleukin-6, vitamin D & diabetes risk-factors modified by a short-term yoga-based lifestyle intervention in overweight/obese individuals. Indian J Med Res. 2015 Jun;141(6):775-82. doi: 10.4103/0971-5916.160698. PMID 26205020